CLINICAL TRIAL: NCT05160077
Title: Noninvasive Characterization of Postprandial Intestinal Blood Flow Using Multispectral Optoacoustic Tomography
Brief Title: Optoacoustic Characterization of Postprandial Intestinal Blood Flow
Acronym: NEPOMUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 346_21 B
Record Dates: First submitted 2021-11-11; First posted 2021-12-16 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2021-11

CONDITIONS: Digestive System Disease; Inflammatory Bowel Diseases
Keywords: optoacoustic; photoacoustic; MSOT; IBD
MeSH Terms: conditions — Digestive System Diseases; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: A comparison is made between 3 study arms:
  A: Fasting,
  B: Standardised breakfast,
  C: Standardised breakfast with added ICG (250mg in 50ml aqua).
  As part of the crossover design, each participant will be assigned to all three study arms on three different days. There is a period of at least 48 hours between two consecutive study days for each subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fasting (Other): All examinations are in a fasting state.
  Interventions: Diagnostic Test: Multispectral optoacoustic tomography (MSOT)
- Standardised Breakfast (Other): Preprandial examination is in fasting state, all postprandial examinations will be conducted with standardized dietary.
  30 minutes after the beginning of the preprandial examination participants receive an standardized breakfast. 270 minutes after the beginning of the preprandial examination participants receive an standardised meal.
  Interventions: Diagnostic Test: Multispectral optoacoustic tomography (MSOT)
- Standardised Breakfast and ICG (Other): Preprandial examination are in a fasting state, all postprandial examinations will be conducted with standardized dietary including indocyanine green (ICG) dye.
  30 minutes after the beginning of the preprandial examination participants receive an standardised breakfast containing ICG. 270 minutes after the beginning of the preprandial examination participants receive an standardised meal without ICG.
  Interventions: Diagnostic Test: Multispectral optoacoustic tomography (MSOT)

INTERVENTIONS:
Diagnostic Test: Multispectral optoacoustic tomography (MSOT) — MSOT Acuity Echo, iThera medical, Munich

SUMMARY:
Inflammatory activities in the gastrointestinal tract are accompanied by an increase in blood flow in the intestinal wall layers of the respective organs. Also in chronic inflammatory bowel diseases, the release of vasoactive inflammatory mediators leads to vasodilation and consecutive increase of blood flow in the bowel wall. So far, these changes in blood flow can be detected by power Doppler sonography without being part of routine clinical diagnostics. Another promising option for non-invasive measurement of blood flow in the intestinal wall is Multispectral Optoacoustic Tomography (MSOT). Previous studies have shown that MSOT can be used to quantitatively measure hemoglobin in the bowel wall and thus provide information on blood flow and inflammatory activity in the intestines of patients with Crohn's disease. This is currently being further investigated in a pivotal study (Euphoria, H2020) and could lead to the possibility of non-invasive assessment of disease activity in inflammatory bowel disease (IBD) in the future.

The regional blood flow in the intestinal wall and the distribution of gastrointestinal blood flow are also subject to strong postprandial changes. During absorption of food components, blood flow increases sequentially in the respective sections of the gastrointestinal tract, leading to postprandial hyperemia. Because postprandial hyperemia is particularly regulated locally by the presence of dietary components, there is a relationship between the sequential increase in blood flow in the intestinal wall and the peristaltic transport of chyme through the gastrointestinal tract. Postprandial hyperemia could also lead to an increase in the optoacoustic hemoglobin signal of the intestinal wall and thus have an impact on the assessment of inflammatory activity in IBD using MSOT. Additionally, MSOT allows the identification of non-absorbable exogenous chromophores, such as indocyanine green (ICG), which could allow co-localization of the chyme in the intestinal lumen after oral application of ICG.

This pilot study investigates whether postprandial blood flow changes can be quantitatively measured using MSOT and whether these changes occur simultaneously with the gastrointestinal passage of the chyme as measured by the ICG signal in the intestinal lumen.

DETAILED DESCRIPTION:
The gastrointestinal tract essentially fulfills two major functions: digestion and absorption of food, and physical and immunological barrier against environmental influences. These basic functions are critically dependent on splanchnic blood flow at both the macrovascular and microvascular levels. In particular, advances in vascular biology have revealed a central and intricate role of blood circulation in inflammatory bowel disease (IBD).

Until now, changes in blood flow have been used as surrogate markers for altered inflammatory activity in the intestine, e.g., by Doppler sonographic detection. Multispectral Optoacoustic Tomograph (MSOT) allows for non-invasive, quantitative imaging of the molecular composition of target tissues. In MSOT, similar to conventional sonography, a transducer is placed on the skin but energy is delivered to the tissue by means of laser light in the near infrared spectrum instead of ultrasound waves. This leads to a constant alternation of minimal expansions and contractions (thermoelastic expansion) of individual tissue components or molecules. The resulting ultrasound waves can subsequently be detected by the same examination unit. Previous studies have shown that quantitative determination of hemoglobin can provide information on blood flow and inflammatory activity in the intestine of adult patients with Crohn's disease. In particular, the distinction between the activity levels of the disease (remission/low/moderate/high) is promising for saving invasive measures in the future when evaluating the progression of the disease.

In addition to inflammatory processes, food intake also causes fluctuations in regional blood flow in the gastrointestinal tract. This manifests as postprandial hyperemia, which occurs sequentially in the different sections of the gastrointestinal tract from oral to aboral.

The time course of postprandial hyperemia in the different sections of the gastrointestinal tract has been scientifically investigated in many studies. While an increase in blood flow in the stomach and duodenum can be detected after 30-60 minutes, it takes much longer for postprandial hyperemia to be detected in the areas used to measure inflammatory activity with MSOT in IBD such as the terminal ileum and sigmoid colon. An increase in blood flow in the ileum can be measured after 120 minutes at the earliest, and the arrival of chyme in the colon and the accompanying local increase in blood flow occur after approximately 240-300 minutes.

It is unclear whether this postprandial hyperemia can lead to a change and potential increase in the optoacoustic hemoglobin signal of the intestinal wall, resulting in falsely high MSOT signals in the determination of inflammatory activity. This study investigates influences of a standardized dietary on the MSOT signal of the intestinal wall using a longitudinal design. Optoacoustic signals will be compared between subjects in fasting and postprandial states. Because the postprandial increase in intestinal blood flow is predominantly a result of the local presence of chyme in the intestine, a simultaneous determination of intestinal transit of chyme during MSOT measurement would be helpful to validate whether postprandial changes in MSOT signals are attributable to hyperemia in the corresponding bowel segment. Besides imaging of hemoglobin, MSOT enables the detection of exogenous chromophores (i.e. dyes). In this study, the oral administration of the nonabsorbable dye indocyanine green (ICG) will be used for noninvasive identification of the chyme. The combination of exogenous and endogenous chromophores thus allows accurate co-localization and registration of intestinal wall blood flow patterns and chyme transit. This information enables accurate anatomical mapping of interfering influences on the determination of hemoglobin using MSOT.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Written declaration of consent

Exclusion Criteria:

Generally valid:

* Pregnancy
* Nursing mothers
* Tattoo in the field of investigation
* Subcutaneous fat tissue over 3 cm
* Chronic or acute diseases of the gastrointestinal tract or symptoms suggestive of such a disease
* Diseases requiring acute treatment
* Lack of written consent

ICG related:

* Known hypersensitivity to ICG, sodium iodide or iodine
* Hyperthyroidism, focal or diffuse thyroid autonomy
* Treatment with radioactive iodine for the diagnostic examination of thyroid function within two weeks before or after the study
* Restricted renal function
* Intake of the following drugs: Beta-blockers, anticonvulsants, cyclopropane, bisulphite compounds, haloperidol, heroin, meperidine, metamizole, methadone, morphine, nitrofurantoin, opium alkaloids, phenobarbital, phenylbutazone, probenecid, rifamycin, any injection containing sodium bisulphite.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Change of the quantitative de-/oxygenated hemoglobin signal (in arbitrary units) | every 60 minutes over 8 hours on each of the three examination days
  Change of the quantitative de-/oxygenated hemoglobin signal in the wall of the gastrointestinal tract (gastric antrum, terminal ileum, transverse colon, and sigmoid colon) over a postprandial time of 7 hours.

SECONDARY OUTCOMES:
Change of the qualitative and quantitative ICG signal (in arbitrary units) | every 60 minutes over 8 hours on on the third examination day
  Change of the qualitative and quantitative ICG signal (in arbitrary units) in the lume of the gastrointestinal tract (gastric antrum, terminal ileum, transverse colon, and sigmoid colon) over a postprandial time of 7 hours.
Change of the quantitative single wavelengths signal (in arbitrary units) | every 60 minutes over 8 hours on each of the three examination days
  Change of the quantitative single wavelengths signal (in arbitrary units) in the wall of the gastrointestinal tract (gastric antrum, terminal ileum, transverse colon, and sigmoid colon) over a postprandial time of 7 hours.
Change of the optoacoustic spectrum (in arbitrary units, normalized) | every 60 minutes over 8 hours on each of the three examination days
  Change of the optoacoustic spectrum (in arbitrary units, normalized) in the wall of the gastrointestinal tract (gastric antrum, terminal ileum, transverse colon, and sigmoid colon) over a postprandial time of 7 hours.
Change of Blood flow in the big splanchnic arteries. | every 60 minutes over 8 hours on each of the three examination days
  Change of Blood flow in the coeliac trunk, superior mesenteric artery, inferior mesenteric artery measured by Doppler sonography over a postprandial time of 7 hours.
Change of Resistance Index in the big splanchnic arteries. | every 60 minutes over 8 hours on each of the three examination days
  Change of Resistance Index in the coeliac trunk, superior mesenteric artery, inferior mesenteric artery measured by Doppler sonography over a postprandial time of 7 hours.
Change of Pulsatility Index in the big splanchnic arteries. | every 60 minutes over 8 hours on each of the three examination days
  Change of Pulsatility Index in the coeliac trunk, superior mesenteric artery, inferior mesenteric artery measured by Doppler sonography over a postprandial time of 7 hours.
Change of peak systolic velocity in the big splanchnic arteries. | every 60 minutes over 8 hours on each of the three examination days
  Change of peak systolic velocity in the coeliac trunk, superior mesenteric artery, inferior mesenteric artery measured by Doppler sonography over a postprandial time of 7 hours.
Change of end diastolic velocity in the big splanchnic arteries. | every 60 minutes over 8 hours on each of the three examination days
  Change of end diastolic velocity in the coeliac trunk, superior mesenteric artery, inferior mesenteric artery measured by Doppler sonography over a postprandial time of 7 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request as follows:
  * Individual participant data will not be available
  * Study Protocol Plan will be available
  * The data will be available beginning 9 months and ending 36 months following article publication.
  * The data will be available to researchers who provide a methodologically sound proposal.
  * The data will be available for individual participant data meta-analysis, only.
  * Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at www.uk-erlangen.de.
  Restrictions may apply due to patient privacy and the General Data Protection Regulation.

REFERENCES:
- [Background] Matheson PJ, Wilson MA, Garrison RN. Regulation of intestinal blood flow. J Surg Res. 2000 Sep;93(1):182-96. doi: 10.1006/jsre.2000.5862. PMID 10945962
- [Background] Deban L, Correale C, Vetrano S, Malesci A, Danese S. Multiple pathogenic roles of microvasculature in inflammatory bowel disease: a Jack of all trades. Am J Pathol. 2008 Jun;172(6):1457-66. doi: 10.2353/ajpath.2008.070593. Epub 2008 May 5. PMID 18458096
- [Background] Calabrese E, Maaser C, Zorzi F, Kannengiesser K, Hanauer SB, Bruining DH, Iacucci M, Maconi G, Novak KL, Panaccione R, Strobel D, Wilson SR, Watanabe M, Pallone F, Ghosh S. Bowel Ultrasonography in the Management of Crohn's Disease. A Review with Recommendations of an International Panel of Experts. Inflamm Bowel Dis. 2016 May;22(5):1168-83. doi: 10.1097/MIB.0000000000000706. PMID 26958988
- [Background] Ntziachristos V, Razansky D. Molecular imaging by means of multispectral optoacoustic tomography (MSOT). Chem Rev. 2010 May 12;110(5):2783-94. doi: 10.1021/cr9002566. No abstract available. PMID 20387910
- [Background] Weber J, Beard PC, Bohndiek SE. Contrast agents for molecular photoacoustic imaging. Nat Methods. 2016 Jul 28;13(8):639-50. doi: 10.1038/nmeth.3929. PMID 27467727
- [Background] Regensburger AP, Brown E, Kronke G, Waldner MJ, Knieling F. Optoacoustic Imaging in Inflammation. Biomedicines. 2021 Apr 28;9(5):483. doi: 10.3390/biomedicines9050483. PMID 33924983
- [Background] Knieling F, Neufert C, Hartmann A, Claussen J, Urich A, Egger C, Vetter M, Fischer S, Pfeifer L, Hagel A, Kielisch C, Gortz RS, Wildner D, Engel M, Rother J, Uter W, Siebler J, Atreya R, Rascher W, Strobel D, Neurath MF, Waldner MJ. Multispectral Optoacoustic Tomography for Assessment of Crohn's Disease Activity. N Engl J Med. 2017 Mar 30;376(13):1292-1294. doi: 10.1056/NEJMc1612455. No abstract available. PMID 28355498
- [Background] Waldner MJ, Knieling F, Egger C, Morscher S, Claussen J, Vetter M, Kielisch C, Fischer S, Pfeifer L, Hagel A, Goertz RS, Wildner D, Atreya R, Strobel D, Neurath MF. Multispectral Optoacoustic Tomography in Crohn's Disease: Noninvasive Imaging of Disease Activity. Gastroenterology. 2016 Aug;151(2):238-40. doi: 10.1053/j.gastro.2016.05.047. Epub 2016 Jun 3. No abstract available. PMID 27269244
- [Background] Goertz RS, Egger C, Neurath MF, Strobel D. Impact of food intake, ultrasound transducer, breathing maneuvers and body position on acoustic radiation force impulse (ARFI) elastometry of the liver. Ultraschall Med. 2012 Aug;33(4):380-5. doi: 10.1055/s-0032-1312816. Epub 2012 Jun 21. PMID 22723037
- [Background] Kvietys PR. The Gastrointestinal Circulation. San Rafael (CA): Morgan & Claypool Life Sciences; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK53092/ PMID 21452437
- [Background] Sou S, Matsui T, Yao T, Naito M, Yorioka M, Beppu T, Nagahama T, Futami K. Differentiating enterocutaneous fistulae from suture abscesses complicating Crohn's disease using oral administration of indocyanine green. J Gastroenterol Hepatol. 2006 Dec;21(12):1850-3. doi: 10.1111/j.1440-1746.2006.04287.x. PMID 17074025
- [Background] Bennink R, Peeters M, Van den Maegdenbergh V, Geypens B, Rutgeerts P, De Roo M, Mortelmans L. Evaluation of small-bowel transit for solid and liquid test meal in healthy men and women. Eur J Nucl Med. 1999 Dec;26(12):1560-6. doi: 10.1007/s002590050495. PMID 10638407
- [Background] Camilleri M, Colemont LJ, Phillips SF, Brown ML, Thomforde GM, Chapman N, Zinsmeister AR. Human gastric emptying and colonic filling of solids characterized by a new method. Am J Physiol. 1989 Aug;257(2 Pt 1):G284-90. doi: 10.1152/ajpgi.1989.257.2.G284. PMID 2764112

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT05160077/Prot_SAP_000.pdf